CLINICAL TRIAL: NCT03012945
Title: Impact of Epidural Anesthesia-analgesia on Long-term Outcome in Elderly Patients After Surgery: 5-year Follow-up of a Multicenter Randomized Controlled Trial
Brief Title: Epidural Anesthesia-analgesia and Long-term Outcome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Peking University First Hospital (Other)
Collaborators: Peking University People's Hospital (Other); Peking University Third Hospital (Other); Beijing Hospital (Other Government); Beijing Shijitan Hospital, Capital Medical University (Other); Peking University (Other)
Responsible Party: Principal Investigator, Dong-Xin Wang, Professor, Peking University First Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: PUCRP201101-1
Record Dates: First submitted 2016-12-31; First posted 2017-01-06 (Estimated); Last update posted 2020-07-08 (Actual); Status verified 2020-07

CONDITIONS: Elderly; Malignant Tumor; Surgical Resection; Epidural Anesthesia; Long-term Outcome
Keywords: Elderly; Cancer surgery; Epidural anesthesia and analgesia; Long-term survival
MeSH Terms: conditions — Neoplasms; Agnosia | interventions — Anesthesia, General

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Combined epidural-general anesthesia (Experimental): Patients assigned to this group (experimental group) receive combined epidural-general anesthesia and postoperative patient-controlled epidural analgesia.
  Interventions: Drug: Combined epidural-general anesthesia
- General anesthesia (Active Comparator): Patients assigned to this group (control group) receive general anesthesia and postoperative patient-controlled intravenous analgesia.
  Interventions: Drug: General anesthesia

INTERVENTIONS:
Drug: Combined epidural-general anesthesia — Combined epidural-general anesthesia and postoperative epidural analgesia. General anesthesia is performed as that in the general anesthesia group. Epidural anesthesia is performed with ropivacaine. Epidural analgesia is performed with a mixture of ropivacaine and sufentanil.
  Other Names: Combined epidural-general anesthesia and postoperative epidural analgesia
  Arms: Combined epidural-general anesthesia
Drug: General anesthesia — General anesthesia and postoperative intravenous analgesia. General anesthesia is performed with propofol induction and propofol and/or sevoflurane maintenance. Intravenous analgesia is performed with morphine.
  Other Names: General anesthesia and postoperative intravenous analgesia
  Arms: General anesthesia

SUMMARY:
Surgical resection is one of the most important treatments for resectable cancer; on the other hand, cancer recurrence and/or metastasis are the major reasons of treatment failure. The development of recurrence/metastasis after cancer surgery mostly depends on the balance between the immunity of human body and the capability of implantation, proliferation and neovascularization of the residual cancer. Preclinical and retrospective clinical studies suggest that anaesthetic management may affect the long-term outcomes after cancer surgery. The investigators hypothesize that use of epidural anesthesia-analgesia may improve long-term survival in elderly patients after major surgery for cancer.

DETAILED DESCRIPTION:
Surgical resection is the main treatment for potentially curable solid organ cancer. However, it is unavoidable that some cancer cells are disseminated into the circulatory or lymphatic system during surgery. And quite a number of patients develop cancer recurrence and/or metastasis after surgery, which are associated with poor long-term outcomes. The development of cancer recurrence and/or metastasis after surgery is mostly dependent on the balance between the anti-tumor immune function of the human body and the ability of implantation, proliferation and neovascularization of the residual cancer cells.

Multiple surgical factors may influence the balance between the anti-cancer immune function and cancer recurrence. For example, the presence of the primary cancer inhibits angiogenesis, whereas cancer resection eliminates this safeguard against angiogenesis; surgical manipulation releases cancer cells into the circulation; surgery-related stress response inhibits natural killer (NK) cell activity and can promote the development of cancer metastasis; local and systemic release of growth factors during surgery may also promote cancer recurrence both locally and at distant sites.

Available studies showed that general anaesthesia/anesthetics may influence the cellular immune function and long-term outcomes. For example, it was found that ketamine and thiopental, but not propofol, suppressed NK cell activity; all three drugs caused a significant reduction in NK cell number; isoflurane and halothane inhibit interferon (IFN) stimulation of NK cell cytotoxicity; nitrous oxide interferes with DNA, purine, and thymidylate synthesis and depresses neutrophil chemotaxis; opioids have been reported to suppress cell-mediated and humoral immunity.

Considering the potential harmful effects of general anesthesia/anesthetics, there is an increasing interest on the effect of regional anaesthesia. Retrospective studies investigating the relationship between epidural anesthesia and outcome after cancer surgery gave different results. In a meta-analysis, regional anesthesia is associated with improved survival (hazard ratio [HR] 0.84, 95% confidence interval [CI] 0.74-0.96, P = 0.013), but not cancer recurrence/metastasis (HR 0.88, 95% Cl 0.64-1.22, P = 0.457). The investigators hypothesize that combined use of epidural anesthesia may produce favorable effects on the long-term survival in elderly patients undergoing major cancer surgery.

ELIGIBILITY:
Inclusion Criteria:

* Elderly patients (age 60-90 years);
* Scheduled to undergo noncardiac thoracic or abdominal surgery with an expected duration of 2 hours or longer. For those who undergo thoracoscopic or laparoscopic surgery, the expected length of incision must be 5 centimeters or more;
* Agree to receive patient-controlled postoperative analgesia.

Exclusion Criteria:

* Refuse to participate;
* Previous history of schizophrenia, epilepsy or Parkinson disease, or unable to complete preoperative assessment due to severe dementia, language barrier or end-stage disease;
* History of myocardial infarction or stroke within 3 months before surgery;
* Presence of any contraindication to epidural anesthesia and analgesia, including abnormal vertebral anatomy, previous spinal trauma or surgery, severe chronic back pain, coagulation disorder (prothrombin time or activated partial prothrombin time longer than 1.5 times of the upper normal limit, or platelet count of less than 80 * 10^9/L), local infection near the site of puncture, and severe sepsis;
* Severe heart dysfunction (New York Heart Association functional classification 3 or above), severe hepatic insufficiency (Child-Pugh grade C), or severe renal insufficiency (serum creatinine of 442 umol/L or above, with or without serum potassium of 6.5 mmol/L or above, or requirement of renal replacement therapy);
* Any other conditions that are considered unsuitable for study participation.

Ages: 60 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1802 (Actual)
Dates: Start 2014-11-01 (Actual); Primary Completion 2019-09-30 (Actual); Study Completion 2019-09-30 (Actual)

PRIMARY OUTCOMES:
Overall survival after surgery. | Up to median 5 years after surgery.
  Time from surgery to the date of all-cause death.

SECONDARY OUTCOMES:
Cancer-specific survival after surgery. | Up to median 5 years after surgery.
  Time from surgery to the date of cancer-specific death. Patients who die from other causes will be censored at the time of death.
Recurrence-free survival after surgery. | Up to median 5 years after surgery.
  Time from surgery to the date of cancer recurrence/metastasis or all-cause death, whichever come first.
Event-free survival after surgery. | Up to median 5 years after surgery.
  Time from surgery to the first date of cancer recurrence/metastasis, new onset cancer, new serious non-cancer disease, or death from any cause.

OTHER OUTCOMES:
Overall survival after surgery (cancer patients). | Up to median 5 years after surgery.
  Time from surgery to the date of all-cause death.
Cancer-specific survival after surgery (cancer patients). | Up to median 5 years after surgery.
  Time from surgery to the date of cancer-specific death. Patients who die from other causes will be censored at the time of death.
Recurrence-free survival after surgery (cancer patients). | Up to median 5 years after surgery.
  Time from surgery to the date of cancer recurrence/metastasis or all-cause death, whichever come first.
Event-free survival after surgery (cancer patients). | Up to median 5 years after surgery.
  Time from surgery to the first date of cancer recurrence/metastasis, new onset cancer, new serious non-cancer disease, or death from any cause.
Cognitive function (3-year survivors). | At the end of the 3rd year after surgery.
  Cognitive function is assessed with the modified Telephone Interview for Cognitive Status (TICS-m; a 12-item questionnaire that assesses global cognitive function by verbal communication via telephone. The score ranges from 0 to 50, with higher score indicating better function).
Quality of life (3-year survivors). | At the end of the 3rd year after surgery.
  Quality of life is assessed with the World Health Organization Quality of Life-brief version (WHOQOL-BREF; a 24-item questionnaire that assesses the quality of life in physical, psychological, social relationship and environmental domains. The score ranges from 0 to 100 for each domain, with higher score indicating better function).

CONTACTS AND LOCATIONS:
Overall Officials: Dong-Xin Wang, MD, Principal Investigator — Peking University First Hospital
Locations (5):
- China (5):
  - Peking University First Hospital, Beijing, Beijing Municipality
  - Beijing Shijitan Hospital, Beijing
  - Peking University People's Hospital, Beijing
  - Peking University Third Hospital, Beijing
  - Beijing Hospital, Beijing

IPD SHARING:
Plan to Share IPD: No
Data will be provided on request.

REFERENCES:
- [Background] Yamaguchi K, Takagi Y, Aoki S, Futamura M, Saji S. Significant detection of circulating cancer cells in the blood by reverse transcriptase-polymerase chain reaction during colorectal cancer resection. Ann Surg. 2000 Jul;232(1):58-65. doi: 10.1097/00000658-200007000-00009. PMID 10862196
- [Background] Shakhar G, Ben-Eliyahu S. Potential prophylactic measures against postoperative immunosuppression: could they reduce recurrence rates in oncological patients? Ann Surg Oncol. 2003 Oct;10(8):972-92. doi: 10.1245/aso.2003.02.007. PMID 14527919
- [Background] Sessler DI. Long-term consequences of anesthetic management. Anesthesiology. 2009 Jul;111(1):1-4. doi: 10.1097/ALN.0b013e3181a913e1. No abstract available. PMID 19512884
- [Background] Buggy DJ, Smith G. Epidural anaesthesia and analgesia: better outcome after major surgery?. Growing evidence suggests so. BMJ. 1999 Aug 28;319(7209):530-1. doi: 10.1136/bmj.319.7209.530. No abstract available. PMID 10463878
- [Background] Melamed R, Bar-Yosef S, Shakhar G, Shakhar K, Ben-Eliyahu S. Suppression of natural killer cell activity and promotion of tumor metastasis by ketamine, thiopental, and halothane, but not by propofol: mediating mechanisms and prophylactic measures. Anesth Analg. 2003 Nov;97(5):1331-1339. doi: 10.1213/01.ANE.0000082995.44040.07. PMID 14570648
- [Background] Mitsuhata H, Shimizu R, Yokoyama MM. Suppressive effects of volatile anesthetics on cytokine release in human peripheral blood mononuclear cells. Int J Immunopharmacol. 1995 Jun;17(6):529-34. doi: 10.1016/0192-0561(95)00026-x. PMID 7499031
- [Background] Markovic SN, Knight PR, Murasko DM. Inhibition of interferon stimulation of natural killer cell activity in mice anesthetized with halothane or isoflurane. Anesthesiology. 1993 Apr;78(4):700-6. doi: 10.1097/00000542-199304000-00013. PMID 8466070
- [Background] Gupta K, Kshirsagar S, Chang L, Schwartz R, Law PY, Yee D, Hebbel RP. Morphine stimulates angiogenesis by activating proangiogenic and survival-promoting signaling and promotes breast tumor growth. Cancer Res. 2002 Aug 1;62(15):4491-8. PMID 12154060
- [Background] Beilin B, Martin FC, Shavit Y, Gale RP, Liebeskind JC. Suppression of natural killer cell activity by high-dose narcotic anesthesia in rats. Brain Behav Immun. 1989 Jun;3(2):129-37. doi: 10.1016/0889-1591(89)90013-5. PMID 2477090
- [Background] Gaspani L, Bianchi M, Limiroli E, Panerai AE, Sacerdote P. The analgesic drug tramadol prevents the effect of surgery on natural killer cell activity and metastatic colonization in rats. J Neuroimmunol. 2002 Aug;129(1-2):18-24. doi: 10.1016/s0165-5728(02)00165-0. PMID 12161016
- [Background] O'Riain SC, Buggy DJ, Kerin MJ, Watson RWG, Moriarty DC. Inhibition of the stress response to breast cancer surgery by regional anesthesia and analgesia does not affect vascular endothelial growth factor and prostaglandin E2. Anesth Analg. 2005 Jan;100(1):244-249. doi: 10.1213/01.ANE.0000143336.37946.7D. PMID 15616085
- [Background] Chen WK, Miao CH. The effect of anesthetic technique on survival in human cancers: a meta-analysis of retrospective and prospective studies. PLoS One. 2013;8(2):e56540. doi: 10.1371/journal.pone.0056540. Epub 2013 Feb 20. PMID 23437162